CLINICAL TRIAL: NCT00183443
Title: Divalproex Extended Release and Placebo, Lithium, or Quetiapine for Mania
Brief Title: Treatment of Mania Symptoms With Drug Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Patricia Suppes, Director, Bipolar and Depression Research Program, National Institute of Mental Health (NIMH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SUP0001AGG/ADO; R01MH069801 (NIH); DSIR 83-ATSO
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-06

CONDITIONS: Bipolar Disorder; Schizophrenia
Keywords: Mania; Manic-depressive; Psychotic disorder
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia; Mania; Psychotic Disorders | interventions — Valproic Acid; Lithium; Lithium Carbonate; Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DVP + placebo (Placebo Comparator): Participants will receive divalproex ER at a therapeutic dose, plus placebo
  Interventions: Drug: Divalproex-extended release (DVP-ER)
- DVP + Quetiapine (Active Comparator): Participants will receive divalproex ER at a therapeutic dose, plus quetiapine up to 800 mg
  Interventions: Drug: Divalproex-extended release (DVP-ER); Drug: Quetiapine
- DVP + Lithium (Active Comparator): Participants will receive divalproex ER at a therapeutic dose, plus lithium at a therapeutic blood level
  Interventions: Drug: Divalproex-extended release (DVP-ER); Drug: Lithium

INTERVENTIONS:
Drug: Divalproex-extended release (DVP-ER) — Divalproex ER will be given in 250 mg or 500 mg tablets. Dosing is once a day, every day, for the duration of study participation, either 12 or 26 weeks.
  Other Names: depakote ER
Drug: Lithium — Extended release lithium will be provided in 300 mg capsules. Participants will be dosed to a therapeutic blood level of lithium from 0.8 to 1.2 mcg/L.
  Other Names: Lithobid
  Arms: DVP + Lithium
Drug: Quetiapine — Quetiapine will be dosed to efficacy, provided in 50 mg, 100 mg, 200 mg, or 300 mg pills.
  Other Names: Seroquel
  Arms: DVP + Quetiapine

SUMMARY:
This study will determine the effectiveness of three different drug therapies in treating the symptoms of mania.

DETAILED DESCRIPTION:
Mania is a serious condition characterized by extreme excitement, mental and physical hyperactivity, insomnia, and disconnected thoughts. Symptoms of mania are common in patients with schizophrenia or bipolar disorder. When associated with these conditions, mania reaches psychotic proportions and often includes hallucinations, paranoia, and feelings of omnipotence. Such symptoms may put individuals with mania and those around them at risk for physical harm. Drug therapies that can safely and effectively treat symptoms of mania are needed. This study will compare three drug combinations in their ability to treat symptoms of mania in people with schizophrenia or bipolar I disorder.

This study will comprise a 12-week acute phase and a 14-week continuation phase. While the acute phase is the primary component of this study, the continuation phase will provide extended data on the characteristics and course of responders to the initial treatment combinations. Results from the continuation phase will be reported elsewhere. In the acute phase, participants will be randomly assigned to receive one of three treatments: divalproex-extended release (DV-ER) and lithium, DV-ER and quetiapine, or DV-ER and placebo. Participants will receive their intervention for 12 weeks. Participants will have weekly study visits for the first 4 weeks of the acute phase; biweekly study visits will occur for the following 8 weeks. After the acute phase, participants who have not responded to their drug regimen will complete their participation in the study.

Participants whose symptoms of mania have decreased will be offered enrollment in the 14-week continuation phase, during which time participants will continue the drug regimen they began in the acute phase. Participants will have biweekly study visits in the continuation phase. During each study visit in both phases, participants will be interviewed about their mania symptoms. Mania, depression, quality of life, and overall functioning scales will assess participants at study entry, at the end of the acute phase, and at the end of the continuation phase. Participants over 50 years of age will have an electrocardiogram (EKG) at study entry to determine cardiac function.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bipolar I disorder or schizophrenia
* Experiencing symptoms of mania at study entry
* Able to speak and understand English
* Willing and able to comply with all study requirements

Exclusion Criteria:

* History of partial response or nonresponse to any of the drugs or drug combinations given in this study
* History of intolerance to DVP, DVP-ER, lithium, or quetiapine
* Disorders that would contraindicate the use of DV, DV-ER, lithium, or quetiapine
* Use of antidepressants within 1 month prior to study entry
* Use of fluoxetine within 3 months prior to study entry
* Impaired cardiac function, as evidenced by abnormal EKG in participants 50 or over
* Unstable medical illness within 2 months prior to study entry
* At risk for suicide
* Substance abuse or dependence within 1 month prior to study entry
* Pregnancy, breastfeeding, or plans to become pregnant during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2005-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trisha Suppes, MD, PhD, Principal Investigator — Stanford School of Medicine and VA Palo Alto Health Care System
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

REFERENCES:
- [Derived] Cosgrove VE, Allende S, Gwizdowski I, Grace Fischer E, Ostacher M, Suppes T. A pilot trial of quetiapine, lithium, or placebo added to divalproex sodium for hypomanic or manic episodes in ambulatory adults with bipolar I disorder. Int J Bipolar Disord. 2022 Mar 2;10(1):7. doi: 10.1186/s40345-022-00252-w. PMID 35235061

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DVP + Placebo | DVP + Quetiapine | DVP + Lithium
Started | 24 | 26 | 25
Completed | 24 (13 eligible participants were offered enrollment in the continuation phase) | 26 (8 eligible participants were offered enrollment in the continuation phase) | 25 (4 eligible participants were offered enrollment in the continuation phase)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DVP + Placebo | DVP + Quetiapine | DVP + Lithium | Total
Number analyzed (Participants) | 24 | 26 | 25 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 26 | 25 | 75
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (11.6) | 33.1 (9.8) | 34.9 (9.0) | 35.6 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 16 | 12 | 38
  Male | 14 | 10 | 13 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 4 | 7
  Not Hispanic or Latino | 22 | 25 | 21 | 68
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 26 | 25 | 75
Mean Number of Lifetime Episodes of Depression [Mean (Standard Deviation); unit: episodes of depression] | 3.4 (1.0) | 3.5 (1.3) | 3.7 (0.9) | 3.5 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Symptoms of Mania, as Measured by Young Mania Rating Scale
Description: Symptoms of mania, as measured by Young Mania Rating Scale. The scale is eleven-item multiple choice diagnostic questionnaire (range 0-60), which psychiatrists use to measure the severity of manic episodes in children and young adults. Typically, 20 is the minimum score required for mania. Higher scores represent increased severity of mania symptoms.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DVP + Placebo | DVP + Quetiapine | DVP + Lithium
Number analyzed (Participants) | 24 | 26 | 25
units on a scale | 5.7 (5.5) | 11.1 (7.8) | 10.0 (6.9)

2. Secondary Outcome: Hamilton Rating Scale for Depression (HAM-D,17)
Description: The Hamilton Rating Scale for Depression is a multiple item questionnaire used to provide an indication of depression, and as a guide to evaluate recovery. The questionnaire is designed for adults and is used to rate the severity of their depression by probing mood, feelings of guilt, suicide ideation, insomnia, agitation or retardation, anxiety, weight loss, and somatic symptoms. The 17-item Likert-type scale (range 0-50) includes eight questions with a 5-point scale (ranging from 0=not present to 4=severe) and nine items scored from 0 to 2. Higher scores indicate increased depression severity. The total sum of these 17 answers is used to arrive at the final score: normal (0-7), mild (8-13), moderate (14-18), severe (19-22), or very severe (>=23).
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DVP + Placebo | DVP + Quetiapine | DVP + Lithium
Number analyzed (Participants) | 24 | 26 | 25
units on a scale | 13.2 (11.6) | 18.3 (9.2) | 18.8 (11.0)

3. Secondary Outcome: Clinical Global Impression Scale for Bipolar Disorder (CGI-BD)
Description: The Clinical Global Impression (CGI) rating scale was modified by Spearing and colleagues (1997) for use in bipolar disorder. CGI scales are measures of symptom severity, treatment response and the efficacy of treatments in treatment studies of patients with mental disorders. The revised CGI-Bipolar Version (CGI-BP) is effective in rating severity of manic and depressive episodes and the degree of change from the immediately preceding phase and from the worst phase of illness. The CGI-BP is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal, not ill) to 7 (very severely ill). Each component of the CGI is rated separately; the instrument does not yield a global score. Only severity of illness scores are reported. Increased scores represent increased illness severity
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DVP + Placebo | DVP + Quetiapine | DVP + Lithium
Number analyzed (Participants) | 24 | 26 | 25
units on a scale | 1.58 (1.02) | 2.54 (1.33) | 2.32 (1.35)

4. Secondary Outcome: Global Assessment of Functioning
Description: The Global Assessment of Functioning (GAF) is a numeric scale used by mental health clinicians and physicians to rate subjectively the social, occupational, and psychological functioning of an individual, e.g., how well one is meeting various problems-in-living. Scores range from 100 (extremely high functioning) to 1 (severely impaired).
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DVP + Placebo | DVP + Quetiapine | DVP + Lithium
Number analyzed (Participants) | 24 | 26 | 25
units on a scale | 68.3 (13.4) | 62.3 (11.1) | 60.8 (10.4)

5. Secondary Outcome: Social and Occupational Functioning Assessment Scale (SOFAS)
Description: The Social and Occupational Functioning Assessment Scale (SOFAS) provides a rating of global social and occupational function independent of clinical symptoms. SOFAS is provided in the Diagnostic and Statistical Manual (DSM-IV) as an Axis V measure. The SOFAS is a global rating of current functioning, which is scored positively on a scale from 0 to 100. Higher scores represent higher levels of functioning. This instrument is a one-item rating of consumer functioning.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DVP + Placebo | DVP + Quetiapine | DVP + Lithium
Number analyzed (Participants) | 24 | 26 | 25
units on a scale | 68.2 (13.7) | 62.1 (11.9) | 59.8 (11.8)

ADVERSE EVENTS:
Arm/Group | DVP + Placebo | DVP + Quetiapine | DVP + Lithium
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 7/24 | 1/26 | 1/25
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DVP + Placebo (N=24) | DVP + Quetiapine (N=26) | DVP + Lithium (N=25)
Increased Appetite (Metabolism and nutrition disorders) | 7 (11) | 1 (12) | 1 (12)
Sedation (General disorders) | 1 (9) | 1 (21) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No